CLINICAL TRIAL: NCT04141696
Title: A Proof-of-Concept Trial on the Effect of Ketamine on Fatigue
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: National Institute of Nursing Research (NINR) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 200003; 20-NR-0003
Record Dates: First submitted 2019-10-25; First posted 2019-10-28 (Actual); Results first posted 2025-04-15 (Actual); Last update posted 2025-04-15 (Actual); Status verified 2025-02-11

CONDITIONS: Fatigue
Keywords: Supportive care; Symptom science; Midazolam; Physiological Effects of Ketamine
MeSH Terms: conditions — Fatigue | interventions — Ketamine; Midazolam

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Ketamine then midazolam administration (Experimental): Participants receive ketamine 0.5 mg/kg intravenous infusion over 40 minutes followed by a two week washout period then receive midazolam 0.045 mg/kg intravenous infusion over 40 minutes followed by two weeks of observation.
  Interventions: Drug: Ketamine; Drug: Midazolam
- Midazolam then ketamine administration (Active Comparator): Participants receive midazolam 0.045 mg/kg intravenous infusion over 40 minutes followed by a two week washout period then receive ketamine 0.5 mg/kg intravenous infusion over 40 minutes followed by two weeks of observation.
  Interventions: Drug: Ketamine; Drug: Midazolam

INTERVENTIONS:
Drug: Ketamine — Given intravenously over 40 minutes
  Other Names: Ketalar
Drug: Midazolam — Used as placebo comparator; given intravenously over 40 minutes
  Other Names: Versed

SUMMARY:
Background:

Many people experience fatigue as a side effect of their illnesses and treatments. There are no medicines to treat fatigue, but a drug called ketamine has reduced fatigue in depressed people. Researchers hope that ketamine, compared to a drug called midazolam, can reduce fatigue in people with illnesses.

Objective:

To test whether ketamine reduces fatigue in cancer survivors and people with chronic illness.

Eligibility:

Adults between the ages of 18 and 70 who have fatigue and are cancer survivors or have been diagnosed with a chronic illness such as chronic fatigue syndrome and lupus.

Design:

Participants will be screened with a physical exam, medical history, blood and urine tests, questions about their fatigue, and breathalyzer test.

During phase 1, participants will complete rating their fatigue using questionnaires. They will be provided thinking, memory, and motivation tests. They will also take a handgrip test. For this study, the participant will have an IV, which a needle guides a thin plastic tube (intravenous or IV line) into an arm in their vein. An IV will be required for two of the visits. They will get a single dose of either ketamine or midazolam through an IV line over 40 minutes. Participants must be accompanied by a responsible friend/family/colleague to take them home after getting the study drug.

Participants will have follow-up visits where they repeat the above tests. They will also have follow-up phone calls.

Phase 2 is the same as phase 1, but participants get the other study drug.

The study lasts 1 month. Each phase lasts 2 weeks. Participants will have 6-8 total NIH visits. For the whole study, they will wear a device on their wrists that records physical activity.

Drug side effects can include vivid dreams, seeing colors, perceiving time as moving slower or faster than normal, dizziness, headache, restlessness, nausea, or vomiting, among others.

DETAILED DESCRIPTION:
Purpose: The purpose of the study is to investigate the anti-fatigue effects of ketamine in individuals with chronic illness.

Background: Although the underlying mechanisms of fatigue have been studied in several disease conditions, the etiology, mechanisms, and risk factors remain elusive and this symptom remains poorly managed. Fatigue is conceptualized as a multidimensional symptom which incorporates temporal, sensory, cognitive/mental, affective/emotional, behavioral, and physiological dimensions. It is described as a common, chronic, and disabling symptom in individuals with Sjogren s syndrome and those with systemic lupus erythematosus. We recently observed that upregulation of glutamate receptors (e.g.,GRM5) can predict individuals who will develop chronic fatigue one year after completing cancer therapy, suggesting that fatigue may share common glutamatergic markers with depression. Ketamine is an N-methyl-D-aspartate (NMDA) receptor antagonist and has been reported to have rapid anti-depressant effects, and we recently found that it also has rapid anti-fatigue effects. Evidence suggest that severe fatigue in diverse medical conditions is driven by similar biological mechanisms, hence identifying a potential anti-fatigue agent in one medical condition may be a valuable anti-fatigue therapy for other fatiguing conditions.

Population for Study: This proof-of-concept study will enroll 59 individuals (target n of completers = 50) with chronic fatigue.

Key Inclusion/Exclusion Criteria: Participants must have a fatigue visual analog scale (VAS) score of greater than or equal to 50 mm (on a 0-100 mm horizontal scale). The greater than or equal to 50 mm fatigue VAS score is considered clinically important fatigue cutoff score for patients with chronic illness, and also captures the effectivity outcome of a previous pharmacologic intervention for fatigue. The participants must not have any progressive or unstable conditions or be taking medications that cause fatigue.

Methodology: This is a phase II, randomized, double-blind (study team and participants), active comparator-controlled, cross-over trial. After determining eligibility during the screening visit, the participant will be randomized to determine the sequence of study drug/active comparator to take during each phase.

Main Study Events / Estimates of Duration and Time Commitments: The study has two periods, and each period is approximately two weeks long (total of four weeks). The study (both periods, excluding the screening visit) will require eight NIH outpatient visits and three phone calls.

Primary and Representative Secondary Outcomes:

* The primary outcome measure of the study is the change in self-reported fatigue visual analogue scale (VAS) score before and three days after receiving ketamine or active comparator (midazolam). A 20% decrease in fatigue VAS score three days after ketamine treatment will be considered the primary indicator of efficacy in this study.
* The secondary outcomes of this study include: physical activity count, skeletal muscle strength, motivation score, cognitive function test scores before and after a dose of ketamine or active comparator.

General Analytic Plans: A linear mixed model with restricted maximum likelihood estimation will be used to examine changes in fatigue symptoms over the course of the trial where all participants with at least a pre-dose and one post-dose measure will be included. Within-subjects factors will include time with pre-dose and all other points. The interaction between time and ketamine treatment will be included along with the fixed intercept. Multiple test corrections (e.g., Bonferroni post hoc tests) will be used to examine differences between levels of significant effects.

ELIGIBILITY:
* INCLUSION CRITERIA:

  1. Have chronic, persistent fatigue for at least 6 months;

     1. Intensity greater than or equal to 50 mm using fatigue VAS (on a 0-100 mm horizontal fatigue scale).
     2. Chronicity greater than or equal to six months total in the past year using the first item of the revised Piper Fatigue Scale.
  2. Be a cancer survivor with a documented medical report of completing primary cancer treatment > 6 months ago (except hormone and vaccine therapies) OR diagnosed with complex syndromes like ME/CFS, CFS, chronic fatigue, fibromyalgia; OR autoimmune disorder such as systemic lupus erythematosus (SLE), or Sjogren s disease;
  3. Able to provide written informed consent;
  4. Able to have an accompanying responsible adult for drug infusion study visits;
  5. 18-70 years of age at the time of signing the informed consent form;
  6. Participants may be NIH employees/staff (see below for some exclusion);
  7. Individuals of childbearing potential must use adequate contraception, as defined below, prior to study entry and for the duration of study participation. Sexually active subjects must agree to use at least one medically accepted barrier method of contraception during the study. For example:

     * Condoms
     * Prescribed hormonal oral contraceptives, vaginal ring, or transdermal patch.
     * Intrauterine device (IUD).
     * Intrauterine hormone-releasing system (IUS).
     * Depot/implantable hormone (e.g., Depo-provera , Implanon).
     * Bilateral tubal occlusion/ligation.
     * Sexual abstinence: refraining from intercourse during the entire period of risk associated with the study requirements or if the participant decides to become sexually active during the study, then one of the highly effective birth control methods must be used.
  8. Individuals of non-childbearing potential; as defined by the following criteria:

     * Postmenopausal defined as 12 months of spontaneous amenorrhea or follicle-stimulating hormone (FSH) serum level > 40 mIU/mL;. appropriate documentation is required.
     * Surgically sterile by hysterectomy and/or bilateral oophorectomy with appropriate documentation of surgical procedure.
     * Has a congenital condition resulting in no uterus. OR
     * Is sterile
     * Has documentation confirming vasectomy

EXCLUSION CRITERIA:

1. Total body irradiation or cranial irradiation for cancer;
2. Has a diagnosis of progressive or unstable disease to any body system causing clinically significant fatigue (e.g., class IV congestive heart failure, end-stage renal disease, liver failure, stage IV chronic obstructive pulmonary disease) including patients with active systemic infections (e.g., human immunodeficiency virus (HIV), active hepatitis, COVID-19 - screened using NIH Clinical Center questionnaire);
3. Individuals with comorbid conditions other than clinically stable cardiovascular, metabolic conditions, and rheumatologic/systemic autoimmune diseases;
4. Current or past psychiatric disorders including medically documented depression with psychosis, bipolar disorder, schizophrenia;
5. Clinically documented post-traumatic stress syndrome and/or traumatic brain injury because of the high risk for ketamine to exacerbate symptoms including hallucinations;
6. Categorized as a high-risk drinker (>=5 drinks/day and >=15 drinks/week for men, >=4 drinks/day and >=8 drinks/week for women). ("Dietary Guidelines for Americans 2015-2020," U.S. Department of Health and Human Services and U.S. Department of Agriculture);
7. Detectable alcohol content >1 mg/dL using either breath test or using other biologic samples (e.g., urine);
8. Current substance use disorder within the last five years as diagnosed on the Structured Clinical Interview for Diagnostic and Statistical Manual (DSM)-5 (SCID-5) or positive urine toxicology results at enrollment;
9. Participants with clinical hypothyroidism or hyperthyroidism defined by abnormal thyroid stimulating hormone (TSH);
10. Poorly controlled hypertension as judged by the Principal Investigator and confirmed by repeat assessment during the screening period (systolic blood pressure (SBP) >160 and diastolic blood pressure (DBP) > 100 in all readings);
11. Any medical condition causing impairment in mobility (e.g., stroke with residual neuromuscular weakness). This may prohibit the assessment of study outcomes, such as physical activity;
12. Any change in dose of regularly scheduled medication or initiation of a new medication (excluding PRN medications) within four weeks prior to signing the informed consent form and throughout the entire duration of the study;
13. Untreated sleep condition.
14. Medically diagnosed kidney disease (except for chronic stable kidney disease with eGFR>45);
15. Medically diagnosed acute narrow-angle glaucoma;
16. Allergic to ketamine, benzodiazepines, flumazenil;
17. With poor IV access;
18. National Institute of Nursing Research (NINR) employees or subordinates, relatives, and/or co-workers of NINR employees/staff or study investigators;
19. Pregnant or lactating individuals;
20. Ongoing medical condition that is deemed by the Principal Investigator to interfere with the conduct or assessments of the study or safety of the participant.
21. Taking concomitant medication known to interact with ketamine and/or midazolam 14 days prior to study drug administration and during the study. The medications are shown in the tables below:

    * List of Psychiatric Medications Allowed and Not Allowed During the Study*

      * Drug Class: Antidepressants;

        * Episodic Use (as needed): No; Chronic Use: No;
        * Restrictions: selective serotonin reuptake inhibitor (SSRI), serotonin-norepinephrine reuptake inhibitors (SNRI), and serotonin modulators, including Bupropion are allowed if on low maintenance doses, and no history of seizure if taking SNRI.
      * Drug class: Antipsychotics;

        --- Episodic Use (as needed): No; Chronic Use: No
      * Drug class: Anxiolytics;

        --- Episodic Use (as needed): No; Chronic Use: No;
      * Drug class: Mood Stabilizers;

        --- Episodic Use (as needed): No; Chronic Use: No;
      * Drug class: Psychotropic drugs not otherwise specified (including herbal products);

        * Episodic Use (as needed): No; Chronic Use: No;
        * Restrictions: No drugs with psychomotor effects or with anxiolytic, stimulant, antipsychotic, or sedative properties are allowed.
      * Drug class: Sedatives/Hypnotics;

        * Episodic Use (as needed): No; Chronic Use: No
    * List of Non-Psychiatric Medications Allowed and Not Allowed During the Study*

      * Drug class: Analgesics;

        * Episodic Use (as needed): Yes; Chronic Use: No;
        * Restrictions: Non-narcotic analgesics only
      * Drug class: Anorexics (sibutramine);

        --- Episodic Use (as needed): No; Chronic Use: No
      * Drug class: Antacids;

        --- Episodic Use (as needed): Yes; Chronic Use: Yes;
      * Drug class: Antianginal Agents;

        --- Episodic Use (as needed): No; Chronic Use: No;
      * Drug class: Antiarrhythmics;

        --- Episodic Use (as needed): No; Chronic Use: No;
      * Drug class: Antiasthma Agents;

        * Episodic Use (as needed): Yes; Chronic Use: Yes
        * Restrictions: Systemic corticosteroids are not allowed if taking more than > 10 mg /day of prednisone or glucocorticoid equivalent.
      * Drug class: Antibiotics;

        * Episodic Use (as needed): Yes; Chronic Use: No;
        * Except erythromycin (see P450-3A4 enzyme inhibitors below)
      * Drug class: Anticholinergics;

        --- Episodic Use (as needed): No; Chronic Use: No;
      * Drug class: Anticoagulants;

        --- Episodic Use (as needed): No; Chronic Use: No;
      * Drug class: Anticonvulsants;

        * Episodic Use (as needed): No; Chronic Use: No;
        * Restrictions: Carbamazepine, phenytoin, and oxcarbazepine are 3A4 inducers and significantly decrease perampanel levels. Topiramate may increase perampanel levels up to 20%
      * Drug class: Antidiarrheal Preparations;

        --- Episodic Use (as needed): Yes; Chronic Use: No;
      * Drug class: Analgesics-Systemic;

        --- Episodic Use (as needed): No; Chronic Use: No;
      * Drug class: Analgesics-Topical;

        --- Episodic Use (as needed): Yes; Chronic Use: Yes;
      * Drug class: Antihistamines-Nonsedating;

        --- Episodic Use (as needed): Yes; Chronic Use: Yes;
      * Drug class: Antihistamines-Sedating;

        --- Episodic Use (as needed): N; Chronic Use: No;
      * Drug class: Antihypertensives;

        * Episodic Use (as needed): Yes; Chronic Use: Yes;
        * Restrictions: Non-narcotic analgesics only
      * Drug class: Anti-inflammatory Drugs;

        * Episodic Use (as needed): Yes; Chronic Use: Yes(a);
        * Restrictions: Systemic corticosteroids are not allowed if taking more than > 10 mg /day of prednisone or glucocorticoid equivalent.
      * Drug class: Antinauseants;

        --- Episodic Use (as needed): Yes; Chronic Use: Yes;
      * Drug class: Antineoplastics;

        * Episodic Use (as needed): No; Chronic Use: No;
        * Restrictions: Agents used in low maintenance doses as immunosuppressive agents (not as antineoplastics) such as Azathioprine, Methotrexate, Mycophenolate mofetil, and Belimumab are allowed.
      * Drug class: Anti-obesity;

        --- Episodic Use (as needed): No; Chronic Use: No;
      * Drug class: Antivirals;

        * Episodic Use (as needed): No; Chronic Use: No;
        * Restrictions: Except for treatment of herpes simplex virus (HSV) with agents without central nervous system (CNS) activity e.g. acyclovir, ganciclovir, famciclovir, valacyclovir
      * Drug class: Cough/Cold Preparations;

        * Episodic Use (as needed): Yes; Chronic Use: No;
        * Restrictions: Dextromethorphan preps- N/N, Guaifenesin - Y/Y, Pseudoephedrine- N/N
      * Drug class: Diuretics;

        * Episodic Use (as needed): Yes; Chronic Use: Yes(b);
        * Restrictions: Non-narcotic analgesics only
      * Drug class: H2-Blockers/ proton pump inhibitor (PPI);

        * Episodic Use (as needed): Yes; Chronic Use: Yes(b);
        * Restrictions: Except cimetidine (see P450-3A4 enzyme inhibitors below)
      * Drug class: Hormones;

        * Episodic Use (as needed): N; Chronic Use: Yes(b);
        * Restrictions: Only thyroid hormone replacement, oral contraceptives, and estrogen replacement therapy are allowed.
      * Drug class: Hypoglycemic Agents;

        * Episodic Use (as needed): No; Chronic Use: Yes(b);
        * Restrictions: Only oral hypoglycemic agents are allowed.
      * Drug class: Antihyperlipidemic

        --- Episodic Use (as needed): No; Chronic Use: No(b);
      * Drug class: Insulin

        --- Episodic Use (as needed): No; Chronic Use: No;
      * Drug class: Laxatives

        --- Episodic Use (as needed): Yes; Chronic Use: Yes;
      * Drug class: Muscle Relaxants

        --- Episodic Use (as needed): No; Chronic Use: No;
      * Drug class: P450-3A4 enzyme inhibitors

        * Episodic Use (as needed): No; Chronic Use: No;
        * Restrictions: Including cimetidine, erythromycin, diltiazem, verapamil, ketoconazole, and itraconazole (topical ketoconazole allowed)
      * Drug class: Protease Inhibitor

        * Episodic Use (as needed): No; Chronic Use: No;
        * Restrictions: Including Saquinavir

a Allowed only if being taken prior to enrolling in the study.

b Allowed only if being taken for at least 2 months prior to enrolling in the study and the dose has been stable for at least 1 month.

*Some medications in the above table may be indicated for exclusionary conditions; therefore, it would be unlikely that participants meeting inclusion will be taking them.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2021-07-26 (Actual); Primary Completion 2024-03-21 (Actual); Study Completion 2024-03-21 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Leorey N Saligan, C.R.N.P., Principal Investigator — National Institute of Nursing Research (NINR)
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: Yes
The datasets generated during and/or analyzed during the current study are available from the corresponding author upon reasonable request.
Time Frame: Publicly available after closure of the study
Access Criteria: De-identified data

REFERENCES:
- [Background] Saligan LN, Luckenbaugh DA, Slonena EE, Machado-Vieira R, Zarate CA Jr. An assessment of the anti-fatigue effects of ketamine from a double-blind, placebo-controlled, crossover study in bipolar disorder. J Affect Disord. 2016 Apr;194:115-9. doi: 10.1016/j.jad.2016.01.009. Epub 2016 Jan 19. PMID 26807672
- [Background] Sharpe M, Wilks D. Fatigue. BMJ. 2002 Aug 31;325(7362):480-3. doi: 10.1136/bmj.325.7362.480. No abstract available. PMID 12202331
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?B_2020-NR-0003.html

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 10 participants were consented and two were screen failure so were not randomized in the study.
Period: Period 1
Arm/Group | Ketamine Then Midazolam Administration | Midazolam Then Ketamine Administration
Started | 4 | 4
Completed | 4 | 4
Not Completed | 0 | 0
Period: Period 2
Arm/Group | Ketamine Then Midazolam Administration | Midazolam Then Ketamine Administration
Started | 4 | 4
Completed | 4 | 4
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- All Study Participants: Participants randomized to receive either ketamine 0.5 mg/kg intravenous infusion over 40 minutes or midazolam 0.045 mg/kg intravenous infusion over 40 minutes followed by a two-week washout period then crossover to receive subsequent treatment followed by two weeks of observation.
Arm/Group | All Study Participants
Number analyzed (Participants) | 8
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 7
  >=65 years | 1
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6
  Male | 2
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 8
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 7
  More than one race | 0
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Percentage Change in Self-reported Fatigue Visual Analog Scale (VAS) Scale
Description: Percentage change in self-reported Fatigue Visual Analog Scale (VAS) after a single intravenous dose of the study drug. The Fatigue VAS is a 0-100 mm scale widely used to assess fatigue in patients with chronic illness. Higher score indicates worse fatigue. Change in fatigue VAS scores measured as comparison of fatigue VAS scores collected at the first visit (baseline) and three days post infusion of study drug during each treatment arm (Ketamine, active comparator). Analysis is measured as the difference between day three score minus the baseline score, divided by the baseline score.
Time Frame: Baseline to three days post infusion for each study arm
Population: All participants who completed the study.
Measure: Median (Inter-Quartile Range); unit: Percentage change
Groups:
- Ketamine Administration: Participants receive ketamine 0.5 mg/kg intravenous infusion over 40 minutes followed by a two week washout period.
- Midazolam Administration: Participants receive midazolam 0.045 mg/kg intravenous infusion over 40 minutes followed by a two week washout period.
Arm/Group | Ketamine Administration | Midazolam Administration
Number analyzed (Participants) | 8 | 8
Percentage change | -21.0 [-28.2 to -7.0] | -12.6 [-27.5 to -6.3]

2. Secondary Outcome: Percentage Change in Self-reported Fatigue Visual Analog Scale (VAS) Scale - Day 7
Description: Percentage change in self-reported Fatigue Visual Analog Scale (VAS) after a single intravenous dose of the study drug. The Fatigue VAS is a 0-100 mm scale widely used to assess fatigue in patients with chronic illness. Higher score indicates worse fatigue. Change in fatigue VAS scores measured as comparison of fatigue VAS scores collected at the first visit (baseline) and seven days post infusion for each treatment arm (Ketamine, active comparator). Analysis is measured as the percentage change in day seven score minus the baseline score, divided by the baseline score.
Time Frame: Up to 7 days post infusion for each study drug
Population: All participants who completed the study.
Measure: Mean (Standard Deviation); unit: Percentage of change
Arm/Group | Ketamine Administration | Midazolam Administration
Number analyzed (Participants) | 8 | 8
Percentage of change | -32.7 (33.9) | -19.6 (22.4)

3. Secondary Outcome: Areas Under the Curve (AUC) for Percentage Changes in Self-reported Fatigue VAS Score - Through Day 7
Description: Percentage change in self-reported Fatigue Visual Analog Scale (VAS) after a single intravenous dose of the study drug. The Fatigue VAS is a 0-100 mm scale widely used to assess fatigue in patients with chronic illness. Higher score indicates worse fatigue. Change in fatigue VAS scores measured as comparison of fatigue VAS scores collected at the first visit (baseline), and then 40, 80, 120, 230 minutes, and 1, 3, and 7 days post infusion for each treatment arm (Ketamine, active comparator). Analysis is measured as the areas under the curve.
Time Frame: Up to 7 days post infusion for each study drug
Population: All participants who completed the study.
Measure: Mean (Standard Deviation); unit: Percentage change*minutes
Arm/Group | Ketamine Administration | Midazolam Administration
Number analyzed (Participants) | 8 | 8
Percentage change*minutes | 497411 (239346) | 518668 (250584)

4. Secondary Outcome: Mean Physical Activity Count Using Actigraphy
Description: Mean physical activity count using actigraphy. Participants wore a portable device to monitor activity levels at day seven post infusion for each study drug. Analysis is measured as the mean of physical activity count on day seven post infusion for each treatment arm.
Time Frame: Day 7 post infusion
Population: All participants who completed the study.
Measure: Mean (Standard Deviation); unit: Count of activity
Arm/Group | Ketamine Administration | Midazolam Administration
Number analyzed (Participants) | 8 | 8
Count of activity | 57.5 (37.0) | 70.4 (35.8)

5. Secondary Outcome: Fatigue Level Measured by Functional Assessment of Chronic Illness Therapy Fatigue (FACIT-F) Scale
Description: The Functional Assessment of Chronic Illness Therapy Fatigue (FACIT-F) Scale is a 13-item questionnaire that measures level of fatigue symptoms. Each item is rated on a scale of 0 (not al all) to 4 (very much) with total score ranging from 0 to 52. Lower score indicates greater fatigue. The Fatigue subscale was used to assess participant's level of fatigue at day seven post infusion for each study arm analyzed as the mean score.
Time Frame: Day 7 post infusion
Population: All participants who completed the study.
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Ketamine Administration | Midazolam Administration
Number analyzed (Participants) | 8 | 8
Units on a scale | 33.8 (6.43) | 33.1 (6.92)

6. Secondary Outcome: Patient Reported Outcome Measurement Information System (PROMIS) - Anxiety Domain
Description: The Patient Reported Outcome Measurement Information System (PROMIS) profile is a self-reported questionnaire assessing quality of life in various domains. The anxiety domain is scored on a 5-point Likert scale and converted into standardized T-scores with a mean of 50 and a standard deviation of 10 based on a US general population. Higher scores indicate more anxiety. Participants completed the computerized adaptive test version of PROMIS anxiety subscale on day seven post infusion and analyzed as mean score.
Time Frame: Day 7 post infusion
Population: All participants who completed the study.
Measure: Mean (Standard Deviation); unit: T Score
Arm/Group | Ketamine Administration | Midazolam Administration
Number analyzed (Participants) | 8 | 8
T Score | 48.0 (10.8) | 48.4 (10.3)

7. Secondary Outcome: Patient Reported Outcome Measurement Information System (PROMIS) - Depression Domain
Description: The Patient Reported Outcome Measurement Information System (PROMIS) profile is a self-reported questionnaire assessing quality of life in various domains. The depression domain is scored on a 5-point Likert scale and converted into standardized T-scores with a mean of 50 and a standard deviation of 10 based on a US general population. Higher score indicates worsening depression. Participants completed the computerized adaptive test version of PROMIS depression subscale on day seven post infusion and analyzed as mean score.
Time Frame: Day 7 post infusion
Population: All participants who completed the study.
Measure: Mean (Standard Deviation); unit: T Score
Arm/Group | Ketamine Administration | Midazolam Administration
Number analyzed (Participants) | 8 | 8
T Score | 45.1 (8.74) | 43.9 (8.76)

8. Secondary Outcome: Patient Reported Outcome Measurement Information System (PROMIS) - Fatigue Domain
Description: The Patient Reported Outcome Measurement Information System (PROMIS) profile is a self-reported questionnaire assessing quality of life in various domains. The fatigue domain is scored on a 5-point Likert scale and converted into standardized T-scores with a mean of 50 and a standard deviation of 10 based on a US general population. Higher score indicates worsening fatigue. Participants completed the computerized adaptive test version of PROMIS fatigue subscale on day seven post infusion and analyzed as mean score.
Time Frame: Day 7 post infusion
Population: All participants who completed the study.
Measure: Mean (Standard Deviation); unit: T Score
Arm/Group | Ketamine Administration | Midazolam Administration
Number analyzed (Participants) | 8 | 8
T Score | 54.0 (6.84) | 54.3 (5.50)

9. Secondary Outcome: Patient Reported Outcome Measurement Information System (PROMIS) - Sleep Disturbance Domain
Description: The Patient Reported Outcome Measurement Information System (PROMIS) profile is a self-reported questionnaire assessing quality of life in various domains. The Sleep Disturbance domain is scored on a 5-point Likert scale and converted into standardized T-scores with a mean of 50 and a standard deviation of 10 based on a US general population. Higher scores indicate worsening sleep disturbance being measured. Participants completed the computerized adaptive test version of PROMIS sleep disturbance subscale on day seven post infusion and analyzed as mean score.
Time Frame: Day 7 post infusion
Population: All participants who completed the study.
Measure: Mean (Standard Deviation); unit: T Score
Arm/Group | Ketamine Administration | Midazolam Administration
Number analyzed (Participants) | 8 | 8
T Score | 52.3 (6.33) | 51.7 (9.28)

10. Secondary Outcome: Fatigue Level Measured by Fatigue Visual Analogue Scale
Description: The fatigue visual analogue scale (VAS) provides a simple method to assess fatigue. The Fatigue VAS is a 0-100 mm scale with 0 (no fatigue at all) to 100 (extreme fatigue). Higher score indicates worsening fatigue. Fatigue VAS score collected from all participants on day seven post infusion for each treatment arm and analyzed as mean score.
Time Frame: Day 7 post infusion
Population: All participants who completed the study.
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Ketamine Administration | Midazolam Administration
Number analyzed (Participants) | 8 | 8
Units on a scale | 45.5 (26.6) | 52.1 (25.8)

11. Secondary Outcome: Measure of Depression Using the Hamilton Rating Scale for Depression (HAM-D)
Description: Hamilton Depression (HAM-D) utilizes a 21-item, clinician-rated paper questionnaire that measures the severity of depressive symptoms of the participants in the past week prior to the interview though only the first 17 items are used in scoring. Depending on the item, it is scored between 0 (not present) and 4 (severe) points using either a three-point or a five-point scale and summed up to obtain the total score. The HAM-D comprises 17 items, of which 9 are evaluated on a five-point scale (0-4) and 8-on a three-point scale (0-2). The total score range from 0 to the maximum score 52 on a 17-item scale, with higher scores indicating more serious depression. Total scores of 0-7 are considered as normal, 8-16 suggest mild depression, 17-23 moderate depression and scores over 24 are indicative of severe depression. Data was collected from all participants on day seven post infusion for each treatment arm and analyzed as mean score.
Time Frame: Day 7 post infusion
Population: All participants who completed the study.
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Ketamine Administration | Midazolam Administration
Number analyzed (Participants) | 8 | 8
Units on a scale | 4.5 (4.04) | 4.5 (4.24)

ADVERSE EVENTS:
Time Frame: Up to 14 days after each infusion intervention
Arm/Group | Ketamine Administration | Midazolam Administration
All-Cause Mortality (participants affected / at risk) | 0/8 | 0/8
Serious Adverse Events (participants affected / at risk) | 0/8 | 0/8
Other Adverse Events (participants affected / at risk) | 8/8 | 8/8
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Ketamine Administration (N=8) | Midazolam Administration (N=8)
Arrhythmia (Cardiac disorders) | 0 | 1
Bradycardia (Cardiac disorders) | 0 | 1
Palpitations (Cardiac disorders) | 1 | 0
Dry mouth (Gastrointestinal disorders) | 2 | 0
Nausea (Gastrointestinal disorders) | 3 | 0
Asthenia (General disorders) | 0 | 2
Anion gap decreased (Investigations) | 1 | 0
Basophil absolute increased (Investigations) | 0 | 1
Basophil count increased (Investigations) | 1 | 1
Blood chloride increased (Investigations) | 1 | 2
Blood creatinine increased (Investigations) | 1 | 1
Blood glucose increased (Investigations) | 4 | 3
Blood pressure increased (Investigations) | 0 | 1
Blood urea increased (Investigations) | 2 | 2
Carbon dioxide increased (Investigations) | 0 | 1
Eosinophil count increased (Investigations) | 0 | 1
Eosinophil percentage decreased (Investigations) | 1 | 1
Eosinophil percentage increased (Investigations) | 0 | 1
Haematocrit decreased (Investigations) | 0 | 1
Haemoglobin decreased (Investigations) | 1 | 1
Immature granulocyte absolute increased (Investigations) | 2 | 3
Immature granulocyte increased (Investigations) | 2 | 5
Lymphocyte absolute decreased (Investigations) | 2 | 2
Lymphocyte percentage increased (Investigations) | 0 | 1
Mean cell haemoglobin concentration decreased (Investigations) | 1 | 1
Mean cell haemoglobin decreased (Investigations) | 1 | 1
Mean cell haemoglobin increased (Investigations) | 1 | 1
Mean cell volume decreased (Investigations) | 1 | 1
Mean platelet volume decreased (Investigations) | 2 | 2
Neutrophil absolute decreased (Investigations) | 0 | 1
Neutrophil absolute increased (Investigations) | 1 | 0
Platelet count decreased (Investigations) | 1 | 1
Platelet count increased (Investigations) | 1 | 1
Red blood cell count decreased (Investigations) | 1 | 1
Red cell distribution width increased (Investigations) | 0 | 1
White blood cell count decreased (Investigations) | 1 | 2
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Dizziness (Nervous system disorders) | 3 | 1
Headache (Nervous system disorders) | 6 | 1
Paraesthesia (Nervous system disorders) | 4 | 2
Presyncope (Nervous system disorders) | 3 | 0
Sensory disturbance (Nervous system disorders) | 1 | 0
Somnolence (Nervous system disorders) | 1 | 1
Vision blurred (Nervous system disorders) | 3 | 0
Dissociation (Psychiatric disorders) | 3 | 0
Dysphoria (Psychiatric disorders) | 2 | 0
Euphoric mood (Psychiatric disorders) | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2024-04-18): https://cdn.clinicaltrials.gov/large-docs/96/NCT04141696/Prot_SAP_000.pdf